CLINICAL TRIAL: NCT06376526
Title: Immuno-consolidation for Newly Diagnosed Multiple Myeloma Using Lack of MRD Negativity After Initial cOmbination Therapy to Pursue Deeper Responses With Linvoseltamab ANd Delay Transplant
Brief Title: IMMUNOPLANT for Newly Diagnosed Multiple Myeloma
Acronym: IMMUNOPLANT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dickran Kazandjian, MD (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Dickran Kazandjian, MD, Professor of Clinical, University of Miami
Organization: University of Miami (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20230236
Record Dates: First submitted 2024-04-16; First posted 2024-04-19 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Linvoseltamab Group (Experimental): Participants in this group will be administered a fixed duration of Linvoseltamab for four to six 28-day cycles, depending on minimal residual disease (MRD) conversion status. After four cycles, participants that are MRD-negative will no longer receive study treatment. Participants that are MRD-positive will receive an additional two cycles of Linvoseltamab.
  Total participation duration is up to 3 years.
  Interventions: Biological: Linvoseltamab

INTERVENTIONS:
Biological: Linvoseltamab — Participants will be administered Linvoseltamab intravenously (IV), using a step-up dosing schedule as follows:
  * Cycle 1, Day 1: 5mg
  * Cycle 1, Day 8: 25mg
  * Cycle 1, Days 15 and 22: 200mg
  * Cycles 2 and 3, Days 1, 8, 15 and 22: 200mg
  * Cycle 4, Days 1 and 15: 200mg.
  For participants who are MRD-positive after four (4) cycles of study treatment:
  * Cycles 5 and 6, Days 1 and 15: 200 mg

SUMMARY:
The purpose of this study is to determine whether Linvoseltamab therapy in patients with newly diagnosed multiple myeloma will convert the disease status from minimal residual disease (MRD)-positive to MRD-negative, and increase the length of time that the disease is controlled. The researchers also want to find out the effects (good and bad) that Linvoseltamab has on participants and the condition.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of newly-diagnosed multiple myeloma (NDMM) per International Myeloma Working Group (IMWG) criteria documented initially prior to induction treatment.
2. Documentation of having received a triplet or quadruplet based initial combination therapy containing at least two of the following: Immunomodulatory drug (IMiD), proteosome inhibitor (PI), and/or anti-cluster of differentiation 38 (anti-CD38).
3. Documentation of attaining a best response of very good partial response (VGPR) or better but MRD+ (sensitivity: ≤10^-5) after at least 4 cycles of combination therapy.

   Note: Patients who at baseline prior to initial combination therapy did not have IMWG evaluable disease and therefore a response assessment of VGPR was unable to be made but currently have residual MM by M-protein and/or involved light chains and/or MRD positivity may enroll. Also, patients who have no apparent bone marrow (BM) residual disease but rather extramedullary disease as evidenced by positron emission tomography (PET)/computed tomography (CT) may enroll.
4. Age ≥18 years.
5. Eastern Cooperative Oncology Group Performance Status (ECOG PS) ≤ 1. Patients with ECOG 2 solely due to local symptoms of myeloma (eg, pain) may be allowed after discussion with the PI (APPENDIX A).
6. Adequate organ function, which is defined as follows:

   * a. Absolute neutrophil count (ANC) ≥1,000 cells/microliter (mcL) (unless patient has ethnic/cyclic neutropenia or if neutropenia is thought to be due to MM)
   * b. Platelets ≥50,000 platelets/mcL
   * c. Hemoglobin ≥8 g/dL (transfusions permitted)
   * d. Serum total bilirubin ≤ 1.5 X upper limit of normal (ULN) or direct bilirubin ≤ ULN for patients with total bilirubin levels > 1.5 ULN (except patients with Gilbert's syndrome who must have a total bilirubin of <3 X ULN)
   * e. Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase (SGOT)) and alanine aminotransferase (ALT) (serum glutamic-pyruvic transaminase (SGPT)) ≤ 2.5 X ULN
   * f. Serum creatinine ≤ 1.5 X ULN (except if due to myeloma) or estimated glomerular filtration rate (eGFR) ≥30 mL/min/1.73 m2 (note that measured glomerular filtration rate [GFR], ie, 24-hour urine, can also be used) based on institutional standard
   * g. Female patients of childbearing potential must have a negative serum pregnancy test at Screening. Female patients of childbearing potential and fertile male patients who are sexually active with a female of childbearing potential must use highly effective methods of contraception throughout the study and for 6 months following the last dose of study treatment. For more information on contraception requirements, please refer to Section 4.11.
   * h. Willing and able to provide written informed consent in accordance with federal, local, and institutional guidelines. The patient must provide informed consent prior to the first screening procedure. For more information on the informed consent process, please refer to Section 15.1.
7. Willing and able to comply with clinic visits and study-related procedures.

Exclusion Criteria:

1. Patients who have received prior systemic therapies for MM other than initial IMiD/PI/anti-CD38-based combination therapy (receiving limited cycles of other induction therapies, eg, cyclophosphamide, bortezomib and dexamethasone (CyBorD) or pulse dexamethasone prior to main induction is allowed). Exclusions include high-dose melphalan with autologous stem cell transplant (HDM-ASCT) and allogeneic stem cell transplant (SCT).

   Note: Continuous systemic corticosteroid treatment with more than 10 mg per day of prednisone or anti-inflammatory equivalent within 72 hours of start of study drug is not permitted.
2. Patients who are receiving any other investigational agents for any reasons.
3. Patients who receive a live attenuated vaccine within 4 weeks of scheduled study treatment administration.
4. Contraindication to any concomitant medication, including those medications administered for infusion reaction, antiviral, antibacterial, anticoagulation, tumor lysis, or hydration prophylaxis given prior to therapy (Sections 4.8, 4.9, and 7).
5. Patient has any of the following:

   1. Human immunodeficiency virus (HIV)-positive with 1 or more of the following:

      * i. History of acquired immune deficiency syndrome (AIDS)-defining conditions cluster of differentiation 4 (CD4) count <350 cells/mm3
      * ii. Detectable viral load during screening or within 6 months prior to screening
      * iii. Not receiving highly active anti-retroviral therapy
      * iv. Had a change in anti-retroviral therapy within 6 months of the start of screening
      * v. Receiving anti-retroviral therapy that may interfere with study treatment as assessed after discussion with the Sponsor-Investigator in consultation with study pharmacist
   2. Hepatitis B infection (ie, hepatitis B surface antigen (HBsAg) or hepatitis B virus (HBV)-deoxyribonucleic acid [DNA] positive). Patients with resolved infection (ie, patients who are HBsAg negative but positive for antibodies to hepatitis B core antigen (anti-HBc) and/or antibodies to hepatitis B surface antigen (anti-HBs)) must be screened using real-time polymerase chain reaction (PCR) measurement of HBV DNA levels. Those who are PCR positive will be excluded. In the event the infection status is unclear, quantitative viral levels are necessary to determine the infection status. EXCEPTION: Patients with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) AND a known history of prior HBV vaccination do not need to be tested for HBV DNA by PCR.
   3. Active hepatitis C infection as measured by positive hepatitis C virus (HCV)-ribonucleic acid (RNA) testing. Participants with a history of HCV antibody positivity must undergo HCV-RNA testing. If a participant with history of chronic hepatitis C infection (defined as both HCV antibody and HCV RNA positive) completed antiviral therapy and has undetectable HCV-RNA 12 weeks following the completion of therapy, the participant is eligible for the study.
6. History of allergic reactions attributed to compounds of similar chemical or biologic composition to the experimental agents used in study.
7. Female patient refuses to discontinue breastfeeding her infant during study treatment or within 6 months after receiving the last dose of study treatment (Section 4.11).
8. Women of childbearing potential (WOCBP) and men who are unwilling to practice highly effective contraception prior to the initial dose/start of the first treatment, during the study, and for at least 6 months after the last dose.

   * Highly effective contraceptive measures for women include: stable use of combined (estrogen and progestogen containing) hormonal contraception (oral, intravaginal, transdermal) or progestogen-only hormonal contraception (oral, injectable, implantable) associated with inhibition of ovulation initiated 2 or more menstrual cycles prior to screening intrauterine device (IUD); intrauterine hormone-releasing system (IUS) bilateral tubal ligation vasectomized partner (provided that the male vasectomized partner is the sole sexual partner of the study participant and that the partner has obtained medical assessment of surgical success for the procedure) and/or sexual abstinence.
   * WOCBP are defined as women who are fertile following menarche until becoming post-menopausal, unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy. A post-menopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient to determine the occurrence of a post-menopausal state.
   * Male study participants with WOCBP partners are required to use condoms unless they are vasectomized or practice sexual abstinence. Male study participants should not donate sperm during the study, and for at least 6 months after the last dose. Vasectomized partner or vasectomized study participant must have received medical assessment of the surgical success.
   * Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient.

   Note: Periodic abstinence (calendar, symptothermal, post-ovulation methods), withdrawal (coitus interruptus), spermicides only, and lactational amenorrhea method (LAM) are not acceptable methods of contraception. Female condom and male condom should not be used together (Section 4.11).
9. Presence of the following cardiac conditions:

   * e. New York Heart Association stage III or IV congestive heart failure
   * f. Myocardial infarction or coronary artery bypass graft ≤ 6 months prior to study enrollment
   * g. History of clinically significant ventricular arrhythmia or unexplained syncope, not believed to be vasovagal in nature or due to dehydration. Uncontrolled cardiac arrhythmia or clinically significant electrocardiogram (ECG) abnormalities
   * h. Unstable or uncontrolled disease/condition related to or affecting cardiac function (eg, unstable angina)
10. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, venous thromboembolic disease, hemorrhage, pulmonary fibrosis, pneumonitis, neurological condition, active autoimmune disease or a documented history of autoimmune disease with the exception of vitiligo, type I diabetes, and prior autoimmune thyroiditis that is currently euthyroid based on clinical symptoms and laboratory testing, or psychiatric illness/social situations within 2 weeks that would limit compliance with study requirements.
11. Active malignancy other than MM requiring treatment in the past 12 months. Malignancies treated within the past 12 months that are considered cured with minimal risk of recurrence are allowed.
12. Have any condition that, in the opinion of the Investigator, would compromise the well-being of the patient or the study or prevent the patient from meeting or performing study requirements.
13. Patients with impaired decision-making capacity will not be enrolled on this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-08-21 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Minimal Residual Disease (MRD) Negativity Rate | Up to 6 months
  The rate of MRD-negativity among participants. Defined by rate of MRD negativity using clonoSEQ MRD® assay at sensitivities of 10^-5 and 10^-6. MRD negativity is defined as 0 residual clonal cells in a bone marrow biopsy sample

SECONDARY OUTCOMES:
Sustained MRD-Negativity Rate | Up to 24 months
  The sustained rate of MRD-negativity among participants will be reported. The duration of time in months measured from the first time the participant achieves an MRD-negative bone marrow (BM) biopsy result until the time the participant has relapsed from MRD-negativity objectively documented with an MRD-positive BM result.
Progression-Free Survival (PFS) | Up to 2 years
  Progression-free survival among study participants will be assessed during treatment and clinical follow-up. PFS is defined as the time from start of treatment until disease progression or death.
Overall Survival | Up to 2 years
  Overall survival (OS) among study participants will be assessed during treatment and clinical follow-up. OS is defined from start of treatment until death from any cause.
Number of Participants Experiencing Treatment-Related Adverse Events | Up to 7 months
  The number of participants experiencing treatment-related adverse events will be reported. Adverse events will be assessed using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Dickran Kazandjian, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No